CLINICAL TRIAL: NCT05139836
Title: Non-Interventional, Prospective Observational Cohort Study to Investigate the Effectiveness and Sustained Disease Control of an Upadacitinib Therapy in Moderate to Severe Atopic Dermatitis Patients Over Two Years
Brief Title: A Study to Assess Disease Activity in Adolescent and Adult Participants With Atopic Dermatitis Who Receive Oral Upadacitinib Tablets in a Real-World Setting
Acronym: UP-TAINED
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P21-705
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis (AD); Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for moderate to severe atopic dermatitis.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Therapies spread over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study will assess the real-world effectiveness of upadacitinib on early and sustained response along adolescent and adult participants with AD. This study also aims to understand upadacitinib utilization patterns in real-world clinical practice.

Upadacitinib (RINVOQ) is approved in the EU for the treatment of moderate to severe AD in adults and adolescents 12 years and older who are candidates for systemic therapy. Approximately 772 adolescent and adult participants with AD will be enrolled at up to 200 sites in Germany.

Participants will receive oral upadacitinib tablets as prescribed by the physician prior to enrolling in this study in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population, and indication. The overall duration of the study is approximately 2 years.

Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=30 kg at baseline for participants between >=12 and <18 years of age.
* Physician confirmed diagnosis of moderate to severe atopic dermatitis at the time of enrollment.
* Upadacitinib initiated as per the local label. The decision to prescribe upadacitinib must have been made prior to and independently of study participation.
* Medical and medication history available at least for the last 6 months.

Exclusion Criteria:

- Current participation in interventional research (note: this does not include non-interventional, post-marketing observational studies, or registry participation).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult participants with atopic dermatitis who have been prescribed upadacitinib in the course of routine practice according to relevant approved licenses.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Disease Control Defined by Atopic Dermatitis Control Tool (ADCT) Total Score <7 Points | Month 3
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percentage of Participants Achieving Disease Control Defined by ADCT Total Score <7 Points Among Participants Who Achieved Disease Control at Month 3 | Month 24
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Disease Control Defined by ADCT Total Score <7 Points | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percentage of Participants with An ADCT Total Score Reduction >=5 from Baseline | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percentage of Participants Achieving Disease Control as Defined by ADCT Item 4 (Sleep Problems) <1 Point and All Other Items <2 Points | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percentage of Participants Achieving Disease Control as Defined by ADCT Total Score <7 Points at Month 3 and Maintaining Disease Control | Up to 21 Months (Excluding Month 3 - Primary Endpoint)
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Absolute Score for ADCT Total Score | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Absolute Change from Baseline for ADCT Total Score | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Time to Achieve ADCT Total Score Reduction >=5 Points from Baseline | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Time to Achieve Disease Control as Defined by ADCT Total Score <7 Points | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percent Change from Baseline for ADCT Total Score | Up to 24 Months
  The ADCT is a validated patient self-administered instrument designed to assess atopic dermatitis (AD) control status in adult and adolescent patients (12 years and older). A higher score indicates lower AD control. A score of >=7 indicates that the patient is not in control.
Percentage of Participants Achieving Eczema Area and Severity Index (EASI) 50 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 75 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 90 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 100 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving Absolute EASI <=7 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Absolute Score for EASI | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Absolute Change from Baseline for EASI | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percent Change from Baseline for EASI | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 50 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 75 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 90 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve EASI 100 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Time to Achieve Absolute EASI <=7 | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 50 in the Head and/or Neck Body Region | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 75 in the Head and/or Neck Body Region | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 90 in the Head and/or Neck Body Region | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving EASI 100 in the Head and/or Neck Body Region | Up to 24 Months
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. The EASI score ranges from 0-72 points with an MCID of 6.6 points. Published score bands: clear (0), almost clear (0.1-1.0), mild AD (1.1-7.0), moderate AD (7.1-21.0), severe AD (21.1-50.0), very severe AD (50.1-72.0).
Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) <=1 | Up to 24 Months
  vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present.) to 4 - Severe (marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
Percentage of Participants Achieving Worst Pruritus Numerical Rating Scale (WP-NRS) <=1 | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving WP-NRS <=3 | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving a WP-NRS Reduction >=4 from Baseline | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Absolute Score for WP-NRS | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Absolute Change from Baseline for WP-NRS | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percent Change from Baseline for WP-NRS | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Time to Achieve WP-NRS <=1 | Up to 24 Months
  WP-NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Absolute Change from Baseline for SCORAD Sleep VAS | Up to 24 Months
  The sleep VAS is one component from the SCORAD test that measures the intensity of sleeplessness during a three day or night recall period. The test uses a VAS scale of 0 to 10 with 0 being "no sleeplessness" and 10 being "worst imaginable sleeplessness".
Absolute Score for Score Atopic Dermatitis (SCORAD) Sleep Visual Analog Scale (VAS) | Up to 24 Months
  The sleep VAS is one component from the SCORAD test that measures the intensity of sleeplessness during a three day or night recall period. The test uses a VAS scale of 0 to 10 with 0 being "no sleeplessness" and 10 being "worst imaginable sleeplessness".
Percent Change from Baseline for SCORAD Sleep VAS | Up to 24 Months
  The sleep VAS is one component from the SCORAD test that measures the intensity of sleeplessness during a three day or night recall period. The test uses a VAS scale of 0 to 10 with 0 being "no sleeplessness" and 10 being "worst imaginable sleeplessness".
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI)/Children's Dermatology Life Quality Index (cDLQI) <=1 | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Percentage of Participants Achieving DLQI/cDLQI <=5 | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Percentage of Participants Achieving DLQI/cDLQI Reduction >=4 from Baseline | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Absolute Score for DLQI/cDLQI | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Absolute Change from Baseline for DLQI/cDLQI | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Percent Change from Baseline for DLQI/cDLQI | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Time to Achieve DLQI/cDLQI <=1 | Up to 24 Months
  DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of subject's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL. For patients from age 12-15 the cDLQI is used.
Absolute Score for Hospital Anxiety and Depression Scale for Anxiety (HADS-A) | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Absolute Change from Baseline for HADS-A | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Percent Change from Baseline for HADS-A | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Absolute Score for Hospital Anxiety and Depression Scale for Depression (HADS-D) | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Absolute Change from Baseline for HADS-D | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Percent Change from Baseline for HADS-D | Up to 24 Months
  The HADS is a 14-item self-report scale, It contains two 7-item scales: one for anxiety (HADS-A) and one for depression (HADS-D). Each HADS item is rated on a 4-point Likert-type scale with total scores on each subscale ranging from 0 to 21, and with higher scores corresponding to greater respective symptom severity.
Absolute Score for Stigmatization (6-Item Stigmatization Scale) | Up to 24 Months
  The scale consists of 6 items that address the feeling of stigmatization because of this condition. The participants respond to each item by 0 (not at all), 1 (sometimes), 2 (very often), or 3 (always). The sum of the responses to the 6 items generates a score ranging from 0 to 18 with higher scores corresponding to a higher feeling of stigmatization.
Absolute Change from Baseline for Stigmatization (6-Item Stigmatization Scale) | Up to 24 Months
  The scale consists of 6 items that address the feeling of stigmatization because of this condition. The participants respond to each item by 0 (not at all), 1 (sometimes), 2 (very often), or 3 (always). The sum of the responses to the 6 items generates a score ranging from 0 to 18 with higher scores corresponding to a higher feeling of stigmatization.
Percent Change from Baseline for Stigmatization (6-Item Stigmatization Scale) | Up to 24 Months
  The scale consists of 6 items that address the feeling of stigmatization because of this condition. The participants respond to each item by 0 (not at all), 1 (sometimes), 2 (very often), or 3 (always). The sum of the responses to the 6 items generates a score ranging from 0 to 18 with higher scores corresponding to a higher feeling of stigmatization.
Absolute Score for Asthma Control Test (ACT) in Participants Having a Confirmed Diagnosis of Asthma at Baseline | Up to 24 Months
  The ACT consists of 5 simple questions regarding the patients' asthma symptom burden. For each question there is a range from 1 to 5. A lower score indicates lower asthma control.
Absolute Change from Baseline in ACT in Participants Having a Confirmed Diagnosis of Asthma at Baseline | Up to 24 Months
  The ACT consists of 5 simple questions regarding the patients' asthma symptom burden. For each question there is a range from 1 to 5. A lower score indicates lower asthma control.
Percent Change from Baseline in ACT in Participants Having a Confirmed Diagnosis of Asthma at Baseline | Up to 24 Months
  The ACT consists of 5 simple questions regarding the patients' asthma symptom burden. For each question there is a range from 1 to 5. A lower score indicates lower asthma control.
Percentage of Participants Achieving Absolute Score >=20 for ACT in Participants Having a Confirmed Diagnosis of Asthma at Baseline | Up to 24 Months
  The ACT consists of 5 simple questions regarding the patients' asthma symptom burden. For each question there is a range from 1 to 5. A lower score indicates lower asthma control.
Percentage of Participants Starting on Upadacitinib 15 mg or 30 mg | Baseline
  Percentage of participants initiating upadacitinib at 15 mg or 30 mg with rationale.
Percentage of Participants with Modification of Upadacitinib Therapy, Timing of Modifications, and Reasons for Modifications | 24 Months
  This includes change in upadacitinib dose with rationale, e.g., dose change, temporary or permanent discontinuation.
Percentage of Participants with Modification of Concomitant AD Therapy, Timing of Modifications, and Reasons for Modifications | 24 Months
  This includes change in concomitant AD therapy with rationale, e.g., adding or removing or changing dose of topical corticosteroids/topical calcineurin inhibitors.
Absolute Score for Skin Pain on the Atopic Dermatitis Symptom Scale (ADerm-SS) | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Percent Change from Baseline for Skin Pain on the ADerm-SS | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Absolute Change from Baseline for Skin Pain on the ADerm-SS | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Absolute Score for Skin Cracking on the ADerm-SS | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Absolute Change from Baseline for Skin Cracking on the ADerm-SS | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Percent Change from Baseline for Skin Cracking on the ADerm-SS | Up to 24 Months
  Skin pain and skin cracking are assessed by a one item test from the ADERM-SS to measure the intensity of skin pain/skin cracking during the past 24 hours. The test uses a scale of 0 to 10, with 0 being "no skin pain"/"no skin cracking" and 10 bring the "worst imaginable skin pain"/"worst imaginable skin cracking".
Absolute Score for Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) of Hand Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Absolute Change from Baseline for vIGA-AD of Hand Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Percent Change from Baseline for vIGA-AD of Hand Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Absolute Score for vIGA-AD of Facial Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Absolute Change from Baseline for vIGA-AD of Facial Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Percent Change from Baseline for vIGA-AD of Facial Eczema | Up to 24 Months
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. It consists of a 5-point scale used by the investigator to measure the severity of disease ranging from 0 - Clear to 4 - Severe.
Absolute Score for Pruritis (5-D Pruritis Scale) | Up to 24 Months
  The 5-D pruritis scale is a brief but multidimensional questionnaire for the quantification of pruritis that is sensitive to change over time. The five dimensions are degree, duration, direction, disability and distribution. The duration, degree and direction domains each include one item, while the disability domain has four items. All items on the first four domains are measured on a five-point Likert scales. The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritis) and 25 (most severe pruritis).
Absolute Change from Baseline for Pruritis (5-D Pruritis Scale) | Up to 24 Months
  The 5-D pruritis scale is a brief but multidimensional questionnaire for the quantification of pruritis that is sensitive to change over time. The five dimensions are degree, duration, direction, disability and distribution. The duration, degree and direction domains each include one item, while the disability domain has four items. All items on the first four domains are measured on a five-point Likert scales. The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritis) and 25 (most severe pruritis).
Percent Change from Baseline for Pruritis (5-D Pruritis Scale) | Up to 24 Months
  The 5-D pruritis scale is a brief but multidimensional questionnaire for the quantification of pruritis that is sensitive to change over time. The five dimensions are degree, duration, direction, disability and distribution. The duration, degree and direction domains each include one item, while the disability domain has four items. All items on the first four domains are measured on a five-point Likert scales. The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritis) and 25 (most severe pruritis).
Absolute Score for Flare Frequency | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. Additionally, the presence of a current flare is assessed at each visit.
Absolute Change from Baseline for Flare Frequency | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. Additionally, the presence of a current flare is assessed at each visit.
Percent Change from Baseline for Flare Frequency | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. Additionally, the presence of a current flare is assessed at each visit.
Absolute Score for Flare Duration | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. The mean duration of the flares is also documented. Additionally, the presence of a current flare is assessed at each visit.
Absolute Change from Baseline for Flare Duration | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. The mean duration of the flares is also documented. Additionally, the presence of a current flare is assessed at each visit.
Percent Change from Baseline for Flare Duration | Up to 24 Months
  Flare frequency is assessed by acquiring information about the number of flares in the last six months before baseline. During the study the patient is asked about number of flares since the last visit. The mean duration of the flares is also documented. Additionally, the presence of a current flare is assessed at each visit.
Absolute Score for Patient Self-Reported Global Assessment of Disease Severity (PtGA) | Up to 24 Months
  Patients assess the overall severity of their disease by a five-point assessment scale (clear, mild, moderate, severe, or very severe, [0-4]), with higher scores corresponding to greater severity.
Absolute Change from Baseline for PtGA | Up to 24 Months
  Patients assess the overall severity of their disease by a five-point assessment scale (clear, mild, moderate, severe, or very severe, [0-4]), with higher scores corresponding to greater severity.
Percent Change from Baseline for PtGA | Up to 24 Months
  Patients assess the overall severity of their disease by a five-point assessment scale (clear, mild, moderate, severe, or very severe, [0-4]), with higher scores corresponding to greater severity.
Percentage of Participants Achieving PtGA <=2 | Up to 24 Months
  Patients assess the overall severity of their disease by a five-point assessment scale (clear, mild, moderate, severe, or very severe, [0-4]), with higher scores corresponding to greater severity.
Percentage of Participants Achieving PtGA Reduction >=1 from Baseline | Up to 24 Months
  Patients assess the overall severity of their disease by a five-point assessment scale (clear, mild, moderate, severe, or very severe, [0-4]), with higher scores corresponding to greater severity.
Incidence and Type of Adverse Events | Up to 24 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug but within 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (125):
- Germany (125):
  - Private Practice - Dr. Sung-Hei Hong-Weldemann /ID# 248844, Freiburg im Breisgau, Baden-Wurttemberg
  - Durani & Durani, Heidelberg,DE /ID# 249172, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinik Heidelberg /ID# 245834, Heidelberg, Baden-Wurttemberg
  - Hautarztpraxis Langenau /ID# 242279, Langenau, Baden-Wurttemberg
  - Flegl MD Stuttgart Germany /ID# 250302, Stuttgart, Baden-Wurttemberg
  - Kurzen, Freising, DE /ID# 241845, Freising, Bavaria
  - Beldio Research GmbH /ID# 245830, Memmingen, Bavaria
  - Dermazent /Id# 268146, Munich, Bavaria
  - Voelkel, Nuremberg, DE /ID# 252445, Nuremberg, Bavaria
  - Hautarzte im Novum Medicum Dr. Kreienkamp & Sautter /ID# 276060, Würzburg, Bavaria
  - Praxis Dres. Freitag/Knoell /ID# 242278, Falkensee, Brandenburg
  - Dermatologie Kleinmachnow /ID# 268383, Kleinmachnow, Brandenburg
  - Praxis Dr. Behnke /ID# 248870, Panketal, Brandenburg
  - Praxis Dr. Asadullah /ID# 243944, Potsdam, Brandenburg
  - Hautärzte am Nauener Tor /ID# 261533, Potsdam, Brandenburg
  - Hautarztpraxis Dr. Alexander Magerl /ID# 270749, Bensheim, Hesse
  - Universitaetsklinikum Frankfurt /ID# 241766, Frankfurt am Main, Hesse
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 243328, Oberursel, Hesse
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 249180, Oberursel, Hesse
  - Hautcentrum Wiesbaden /ID# 274848, Wiesbaden, Hesse
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 241658, Bramsche, Lower Saxony
  - Praxis Dres. Kaspari /Schenck /ID# 241688, Hanover, Lower Saxony
  - Herrmann, Greifswald, DE /ID# 241889, Greifswald, Mecklenburg-Vorpommern
  - Hoeller-Obrigkeit, Aachen, DE /ID# 245430, Aachen, North Rhine-Westphalia
  - Klinikum Rosenhoehe /ID# 241601, Bielefeld, North Rhine-Westphalia
  - Katholisches Klinikum Bochum gGmbH /ID# 270537, Bochum, North Rhine-Westphalia
  - Kramer/Mortazawi, Remscheid /ID# 241824, Remscheid, North Rhine-Westphalia
  - Karl, Soest, DE /ID# 241909, Soest, North Rhine-Westphalia
  - Bell, Andernach, DE /ID# 249154, Andernach, Rhineland-Palatinate
  - Grossmann, Koblenz, DE /ID# 242992, Koblenz, Rhineland-Palatinate
  - Hautarztpraxis Dr. Kirschner /ID# 266738, Mainz, Rhineland-Palatinate
  - CMS3 Company for Medical Study /ID# 241659, Selters, Rhineland-Palatinate
  - Dermatologisches Studienzentrum am Haut- und Laserzentrum /ID# 243882, Simmern, Rhineland-Palatinate
  - HMS GmbH Zimmer /ID# 241657, Merzig, Saarland
  - Praxis P. Hausler-Mehlhorn /ID# 241527, Chemnitz, Saxony
  - Neubauer, Leipzig, DE /ID# 241823, Leipzig, Saxony
  - Praxis Dr. Raschke /ID# 251398, Magdeburg, Saxony-Anhalt
  - Praxis Dr. Mempel /ID# 241827, Elmshorn, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 240096, Kiel, Schleswig-Holstein
  - Dermatologie Moelln Praxis Dr. Bodo Segert /ID# 242280, Mölln, Schleswig-Holstein
  - Praxis Liebetrau /ID# 271896, Friedrichroda, Thuringia
  - Petri, Ahaus, DE /ID# 243452, Ahaus
  - Dr. Stoeber /ID# 251066, Ahlen
  - Praxis Dr. Mihaescu /ID# 241825, Augsburg
  - MVZ medicum.mittelhessen /ID# 266126, Bad Camberg
  - Mauer, Bad Kreuznach, DE /ID# 241990, Bad Kreuznach
  - Timmel/Timm/Vorwerk, Bergen /ID# 241661, Bergen
  - Hautarztpraxis Dr. med. Christiane Handrick /ID# 262667, Berlin
  - Praxis Dermatologie am Savigny /ID# 248846, Berlin
  - Private Practice - Dr. Gellrich, Dr. Klein & Dr. Soost /ID# 250301, Berlin
  - Schirmer, Berlin, DE /ID# 241684, Berlin
  - Kors, Berlin, DE /ID# 241847, Berlin
  - Dues/Manasterski, Berlin, DE /ID# 243885, Berlin
  - Hautarztzentrum Tegel /ID# 241826, Berlin
  - Haut Pur - Dermatologische Gemeinschaftspraxis /ID# 243943, Berlin
  - Hautarztpraxis Dr. Weid /ID# 265213, Bingen am Rhein
  - Praxis fuer Innere Medizin/Rheumatologie /ID# 241846, Blaubeuren Abbey
  - Praxis T. Schadeck /ID# 241768, Bogen
  - Barth, Borna, DE /ID# 248871, Borna
  - Schwichtenberg, Bremen, DE /ID# 241683, Bremen
  - Dr. Hoffmann /ID# 245423, Cologne
  - Derma Köln /ID# 241856, Cologne
  - Praxis Dr. Sbornik /ID# 241818, Deggendorf
  - Hautmedizin Delitzsch /ID# 251394, Delitzsch
  - Richter-Huhn, Dresden, DE /ID# 241822, Dresden
  - Praxis Dr. Korge /ID# 241531, Düren
  - Hautarztpraxis Friedberg Dr. med. Wilfried Jungkunz /ID# 248851, Friedberg (Hessen)
  - Rotterdam, Gelsenkirchen, DE /ID# 241819, Gelsenkirchen
  - Gemeinschaftspraxis Rietkoetter und Jablonka /ID# 241821, Gelsenkirchen
  - Praxis Dr. Lange /ID# 241829, Gera
  - Loth, Gernsbach, DE /ID# 241828, Gernsbach
  - Hautarztpraxis Dr. Budihardja /ID# 241851, Giessen
  - Brinkmann & Partner, Gladbeck, /ID# 241850, Gladbeck
  - Dr. Krueger /ID# 265150, Goslar
  - Grossmann, Grossenhain, DE /ID# 250303, Großenhain
  - Praxis Dr. Wegener /ID# 263731, Hamburg
  - Cutaneum /ID# 249104, Hamburg
  - Dermatologikum Hamburg /ID# 245431, Hamburg
  - Duplicate_Hautarztpraxis Luetten/Sack /ID# 241534, Hamburg
  - Dr. Wrage-Brors /ID# 262705, Hamburg
  - Mensing Derma MVZ GmbH /ID# 272383, Hamburg
  - Private Practice - Dr. Daniela Kasche - Langelohstrasse /ID# 249102, Hamburg
  - MVZ Prof. Dr. Ockenfels Haut- und Allergie-Praxisklinik GmbH /ID# 245395, Hanau
  - Dr. Buerkle /ID# 250299, Haslach im Kinzigtal
  - Hautarztpraxis Haßberge /ID# 257648, Haßfurt
  - Gemeinschaftspraxis Dres. Anika Hünermund/Mario Pawlak /ID# 241908, Heilbad Heiligenstadt
  - Haut- u. Laserzentrum Heilbronn /ID# 250305, Heilbronn
  - Hausarztpraxis & Laserzentrum Dr. Zimmermann & Kollegen /ID# 251051, Heusenstamm
  - Praxis Dres. Bischoff/Danz /ID# 241852, Ilmenau
  - Stockmeier, Ingoldstadt, DE /ID# 248877, Ingolstadt
  - Hautarztpraxis Weidgang /ID# 248850, Jülich
  - Derma Sana /ID# 241854, Karlsruhe
  - Dermatologische Praxis Kempen /ID# 248852, Kempen
  - Praxis Dres. Bornemann/Reinerth /ID# 257649, Krefeld
  - Dres. Jacobs & Kollegen /ID# 241989, Kulmbach
  - Praxis Dres. Wiemers/Wiemers /ID# 241602, Leipzig
  - Haut- und Allergie-Zentrum Lippstadt /ID# 241929, Lippstadt
  - Hagemeier, Loehne, DE /ID# 241886, Löhne
  - Magdeburger Company for Medical Studies & Services GmbH /ID# 248849, Magdeburg
  - MVZ "Im Altstadtquartier" Magdeburg /ID# 261366, Magdeburg
  - Universitaetsklinikum Magdeburg /ID# 249174, Magdeburg
  - Hausärzte am Fastnachtsbrunnen /ID# 250304, Mainz
  - Dermatologie Quist-BAG Dres. med. Quist PartG /ID# 243325, Mainz
  - Praxis A. Viculova /ID# 266133, Miltenberg
  - ZENTderma /ID# 241539, Mönchengladbach
  - Dermatologie im Tal Praxis Dr.med. Maria Leibl /ID# 266128, Munich
  - Hautzentrum am Marienplatz /ID# 248847, Munich
  - Quack, Munich, DE /ID# 241536, Munich
  - Dr. Gißler-Walter /ID# 248876, Mutterstadt
  - Dr. Rezai /ID# 250298, Münster
  - Dermatologie im Apfelgarten /ID# 263704, Neu Wulmstorf
  - Praxis Dr. Konstantin Ertner /ID# 249153, Nuremberg
  - Hockmann, Oelde, DE /ID# 241906, Oelde
  - Harzklinikum Dorothea Christiane Erxleben /ID# 251067, Quedlinburg
  - Dr. Schaefers /ID# 255492, Reutlingen
  - Praxis Dr. Fränken /ID# 241853, Schwelm
  - Gemeinschaftspraxis fur Dermatologie /ID# 245831, Stadtroda
  - Praxis Dr. Termeer /ID# 241662, Stuttgart
  - Jasnoch/Kock/Borrosch, Vechta, /ID# 252081, Vechta
  - Barnikol, Waltershausen, DE /ID# 241844, Waltershausen
  - Praxis Dehmel / Brand-Opitzer /ID# 243884, Wasserburg A. Inn
  - Dr. Barbara Kempkes, Werne /ID# 241910, Werne
  - Dr. med. Nicola Möller & Thomas Kurtenbach GbR Dermatologie im Zentrum /ID# 266130, Wiesbaden
  - Hautarztpraxis Dr. med. Matthias Hoffmann /ID# 241907, Witten
  - Albrecht, Wurzen, DE /ID# 241988, Wurzen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weidinger S, Schadeck T, Jacobs F, Weyergraf A, Mortazawi D, Hagemann T, Abousamra F, Mosch T, Fritz B, Lauffer F. Early Achievement of High Treatment Targets in Moderate-to-Severe Atopic Dermatitis with Upadacitinib: Real-World Evidence from the Observational UP-TAINED Study. Dermatol Ther (Heidelb). 2025 Apr;15(4):919-931. doi: 10.1007/s13555-025-01373-7. Epub 2025 Mar 15. PMID 40087231
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/